CLINICAL TRIAL: NCT02151344
Title: Phase 1 Evaluation of the Optimal Interval Between Priming With a Live Influenza A Vaccine H7N9 (6-2) AA ca Recombinant (A/Anhui/1/2013 (H7N9) x A/Ann Arbor/6/60 ca), a Live Attenuated Virus Vaccine Candidate for Prevention of Influenza H7N9 Disease Followed by Boost With a Non-adjuvanted Inactivated H7N9 Influenza Vaccine
Brief Title: Evaluating the Safety and Immune Response to a Live H7N9 Influenza Virus Vaccine Followed by an Inactivated H7N9 Influenza Virus Vaccine, Given at Varying Intervals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CIR 293
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Influenza A Virus, H7N9 Subtype

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 (Experimental): Participants will receive one dose of the H7N9 A/Anhui/13 ca influenza virus vaccine at Day 0 and one dose at Day 28. They will then receive one dose of the inactivated subvirion H7N9 vaccine 1 month later.
  Interventions: Biological: H7N9 A/Anhui/13 ca influenza virus vaccine; Biological: Inactivated subvirion H7N9 vaccine
- Cohort 2 (Experimental): Participants will receive one dose of the H7N9 A/Anhui/13 ca influenza virus vaccine at Day 0 and one dose at Day 28. They will then receive one dose of the inactivated subvirion H7N9 vaccine 2 months later.
  Interventions: Biological: H7N9 A/Anhui/13 ca influenza virus vaccine; Biological: Inactivated subvirion H7N9 vaccine
- Cohort 3 (Experimental): Participants will receive one dose of the H7N9 A/Anhui/13 ca influenza virus vaccine at Day 0. They will then receive one dose of the inactivated subvirion H7N9 vaccine 2 months later.
  Interventions: Biological: H7N9 A/Anhui/13 ca influenza virus vaccine; Biological: Inactivated subvirion H7N9 vaccine
- Cohort 4 (Experimental): Participants will receive one dose of the H7N9 A/Anhui/13 ca influenza virus vaccine at Day 0. They will then receive one dose of the inactivated subvirion H7N9 vaccine 1 month later.
  Interventions: Biological: H7N9 A/Anhui/13 ca influenza virus vaccine; Biological: Inactivated subvirion H7N9 vaccine
- Cohort 5 (Experimental): Participants will receive one dose of the inactivated subvirion H7N9 vaccine at Day 0 and one dose at Day 28.
  Interventions: Biological: Inactivated subvirion H7N9 vaccine

INTERVENTIONS:
Biological: H7N9 A/Anhui/13 ca influenza virus vaccine — Participants will receive approximately 10^7.0 fluorescent focus units (FFU) of the vaccine; the vaccine will be administered with a nose spray device.
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Biological: Inactivated subvirion H7N9 vaccine — Participants will receive a dose of 30 mcg of the vaccine; the vaccine will be administered as an injection.

SUMMARY:
H7N9 viruses have caused a recent outbreak of severe illness in humans in China. The purpose of this study is to evaluate the safety and immune response of an H7N9 A/Anhui/13 ca influenza virus vaccine followed by an inactivated subvirion H7N9 vaccine at varying intervals.

DETAILED DESCRIPTION:
H7N9 avian influenza (AI) viruses have been responsible for a recent outbreak of illness in humans in China, which was associated with severe respiratory illnesses resulting in acute respiratory distress syndrome (ARDS) and intensive care unit (ICU) admissions. The purpose of this study is to evaluate the safety, infectivity, and immunogenicity of a live attenuated H7N9 A/Anhui/13 cold adapted (ca) influenza virus vaccine followed by a boost with an inactivated subvirion H7N9 vaccine at varying intervals.

This study will enroll participants into five cohorts. Participants in Cohorts 1, 2, 3, and 4 will be admitted to an isolation unit on Study Day -2. On Study Day 0, participants will receive one dose of the H7N9 A/Anhui/13 ca influenza virus vaccine via a nose spray device. While in the isolation unit, participants will undergo a physical examination and nasal wash each day, and a blood collection on select days. Participants will remain in the isolation unit for at least 9 days after receiving the vaccine, but possibly longer, depending on their test results.

Participants in Cohorts 1 and 2 will return to the isolation unit 4 to 8 weeks after receiving the first vaccine (at approximately Day 28). They will receive the second dose of the H7N9 A/Anhui/13 ca influenza virus vaccine and repeat all of the same procedures that occurred after the first vaccination.

Participants will then receive one dose of the inactivated subvirion H7N9 vaccine 1 month (Cohort 1) or 2 months (Cohort 2) after receiving the second vaccine.

Participants in Cohorts 3 and 4 will receive the inactivated subvirion H7N9 vaccine either 1 month (Cohort 4) or 2 months (Cohort 3) after receiving one dose of the live attenuated vaccine. For Cohorts 1-4, participants study visits will occur 7, 14, 28, and 90 days after receiving the vaccine and will include a medical history review, physical examination, and blood collection at select visits.

Participants in Cohort 5 will receive one dose of the inactivated subvirion H7N9 vaccine at Day 0 and one dose at Day 28. Study visits will occur on Days 0, 7, 28, 35, 42, 56, and 118, and will include blood collections and physical examinations. Participants in Cohort 5 will not be admitted to the isolation unit.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and non-pregnant females between 18 years and 49 years of age, inclusive. Children will not be recruited or enrolled in this study because they are not in the apparent risk group, for safety considerations, and because of the need for isolation.
* General good health, without significant medical illness, physical examination findings, or significant laboratory abnormalities as determined by the investigator
* Agree to storage of blood specimens for future research
* Available for the duration of the trial
* Willingness to participate in the study as evidenced by signing the informed consent document
* Female participants of childbearing potential must agree to use effective birth control methods for the duration of the study (for example, pharmacologic contraceptives including oral, parenteral, and transcutaneous delivery; condoms with spermicide; diaphragm with spermicide; intrauterine device; abstinence from heterosexual intercourse; surgical sterilization). All female participants will be considered being of childbearing potential except those who have undergone hysterectomy and those in whom menopause occurred at least 1 year prior to the study.

Exclusion Criteria:

* Pregnancy, as determined by a positive human choriogonadotropin (beta-HCG) test
* Currently breastfeeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies including urine testing
* Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the study protocol
* Previous enrollment in an H7 influenza vaccine trial or in any study of an avian influenza vaccine
* Seropositive to the H7N9 influenza A virus (serum HAI titer greater than 1:8)
* Positive urine drug toxicology test indicating narcotic use/dependency
* Have medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* History of anaphylaxis
* Allergy to oseltamivir as determined by participant report
* Current diagnosis of asthma or reactive airway disease (within the past 2 years)
* History of Guillain-Barré Syndrome
* Positive enzyme-linked immunosorbent assay (ELISA) and confirmatory test (e.g., Western blot or HIV-1/HIV-2 differentiation assay) for human immunodeficiency virus-1 (HIV-1)
* Positive ELISA and confirmatory test (e.g., recombinant immunoblot assay) for hepatitis C virus (HCV)
* Positive hepatitis B virus surface antigen (HBsAg) by ELISA
* Known immunodeficiency syndrome
* Use of corticosteroids (excluding topical preparations) or immunosuppressive drugs within 30 days prior to vaccination
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to study vaccination
* History of asplenia
* Body mass index (BMI) greater than 40
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study vaccination
* Current smoker unwilling to stop smoking for the duration of the study. More information on this criterion is available in the protocol.
* Travel to the Southern Hemisphere within 14 days prior to study vaccination
* Travel on a cruise ship within 14 days prior to study vaccination
* Receipt of another investigational vaccine or drug within 30 days prior to study vaccination
* History of hypersensitivity to any component of the investigational product including egg or egg protein, or serious, life threatening, or severe reactions to previous influenza vaccinations
* Individuals who use intranasal medications chronically
* Receipt of antiviral therapy or antiviral agents within 48 hours prior to receipt of investigational product

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Measurement of the ability of the pLAIV vaccine to induce priming by assessing the response to a subsequent dose of pIIV | Measured through participants' last study visit: 90 days after receiving the last vaccine (Cohorts 1-4) or Day 118 (Cohort 5)
Measurement of the optimal interval between the priming with pLAIV and the subsequent boost with pIIV | Measured through participants' last study visit: 90 days after receiving the last vaccine (Cohorts 1-4) or Day 118 (Cohort 5)
Determination of whether 1 dose or 2 doses of pLAIV followed by a pIIV boost is sufficient to induce an optimal immune response | Measured through participants' last study visit: 90 days after receiving the last vaccine (Cohorts 1-4) or Day 118 (Cohort 5)
Frequency of vaccine-related reactogenicity events (REs) for 2 doses of pLAIV vaccine followed by a single dose of inactivated pIIV and compare to 2 doses of pIIV alone | Measured through participants' last study visit: 90 days after receiving the last vaccine (Cohorts 1-4) or Day 118 (Cohort 5)
Frequency of other adverse events (AEs) for 2 doses of pLAIV vaccine followed by a single dose of inactivated pIIV and compare to 2 doses of pIIV alone | Measured through participants' last study visit: 90 days after receiving the last vaccine (Cohorts 1-4) or Day 118 (Cohort 5)

SECONDARY OUTCOMES:
Number of vaccinees infected with the H7N9 Anhui 2013/AA ca recombinant vaccine candidate | Measured through participants' last study visit: 90 days after receiving the last vaccine (Cohorts 1-4) or Day 118 (Cohort 5)
  Infection is defined as recovery of vaccine virus from nasal wash, detection of virus in nasal wash by rRT-PCR, and/or a greater than or equal to 4-fold rise in antibody titer.
Measurement of the amount of vaccine virus shed by each recipient | Measured through participants' last study visit: 90 days after receiving the last vaccine (Cohorts 1-4) or Day 118 (Cohort 5)
Measurement of amount of serum and nasal wash antibody induced by the vaccine | Measured through participants' last study visit: 90 days after receiving the last vaccine (Cohorts 1-4) or Day 118 (Cohort 5)
Capacity of the H7N9 Anhui 2013/AA ca recombinant vaccine candidate to elicit HAI and neutralizing antibodies to future H7 influenza viruses | Measured through participants' last study visit: 90 days after receiving the last vaccine (Cohorts 1-4) or Day 118 (Cohort 5)
  Includes the development of a serum bank

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar Talaat, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States